CLINICAL TRIAL: NCT03804515
Title: A Phase 1 Study for the Evaluation of Excretion (Mass Balance) and Pharmacokinetics of 14C-Labeled Poziotinib in Cancer Patients Suitable for Treatment With Poziotinib
Brief Title: A Mass Balance and Pharmacokinetics Study of 14C-Labeled Poziotinib in Cancer Patients Suitable for Treatment With Poziotinib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-102
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Solid Tumor
Keywords: EGFR; HER2 mutations; EGFR/HER2 overexpression/amplification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C-labeled Poziotinib (Experimental)
  Interventions: Drug: 14C-labeled poziotinib

INTERVENTIONS:
Drug: 14C-labeled poziotinib — a single capsule containing 12 mg of 14C-labeled poziotinib (approximately 90 to 110 μCi) will be administered orally

SUMMARY:
The purpose of this study is to determine routes of excretion and single-dose PK parameters for poziotinib in patients with solid tumors with EGFR or HER2 mutations or EGFR/HER2 overexpression/amplification.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose study of 14C-labeled poziotinib to determine routes of excretion and single-dose PK parameters for poziotinib in patients with solid tumors with EGFR or HER2 mutations or EGFR/HER2 overexpression/amplification.

On Day 1, enrolled patients will be admitted to the inpatient unit and all predose assessments will be completed. Patients will be admitted to the inpatient unit for 9 days. On Day 2, a single capsule containing 12 mg of 14C-labeled poziotinib (approximately 90 to 110 μCi) will be administered orally in the morning right after breakfast with at least 200 mL of water.

Over the following 168 hours, urine and feces will be collected and pooled at specified intervals for measurement of total radioactivity recovered and subsequent determination of the routes of elimination of poziotinib and its metabolites. Blood samples will be taken at specified time points for 168 hours after dosing for estimation of single-dose poziotinib PK parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient can be male or female and is at least 18 years of age
* Patient must be willing and capable of giving written Informed Consent and willing to stay in the research unit for 9 days.
* Patient has a life expectancy of at least 6 months.
* Histological confirmation of solid tumor cancer that is suitable for poziotinib therapy. These may include patients with any solid malignancy with either EGFR or HER 2 mutations or EGFR/HER2 overexpression/amplification. Brain metastases are allowed, if patient is clinically stable and does not require treatment with anticonvulsants or escalating steroid doses.

Exclusion Criteria:

* Patient has a diagnosis of primary and or metastatic hepatic or renal carcinomas.
* Patient is unable to take oral medication or has ongoing Grade ≥2 diarrhea due to any etiology including Crohn's disease and/or ulcerative colitis.
* Previous poziotinib exposure
* Patient has previously participated in a study utilizing 14C.
* Patient has any pathology or history of procedures expected to change absorption
* Patient has a PEG (Percutaneous Endoscopic Gastrostomy) tube

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Maximum recovery of the radioactive dose in plasma, urine and feces | 1 year
  The route of excretion of radioactive poziotinib and its metabolites following single oral administration of 14C-labeled poziotinib in patients with solid tumors suitable for treatment with poziotinib.

SECONDARY OUTCOMES:
The concentration of 14C-labeled poziotinib and its metabolites in plasma, urine and feces | 1 year
  To identify major metabolites of poziotinib

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States